CLINICAL TRIAL: NCT04474470
Title: A Phase 1/2 Study with Open-Label, Dose Escalation Phase Followed by Single-Arm Expansion At the Maximum Tolerated Dose to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of NT219 Injection Alone and in Combination with ERBITUX® (Cetuximab) in Adults with Advanced Solid Tumors and Head and Neck Cancer
Brief Title: A Study to Evaluate NT219 Alone and in Combination with ERBITUX® (Cetuximab) in Adults with Advanced Solid Tumors and Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TyrNovo Ltd. (Industry)
Responsible Party: Sponsor
Organization: Purple Biotech Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYR-219-01
Record Dates: First submitted 2020-06-30; First posted 2020-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor, Adult; Squamous Cell Carcinoma of Head and Neck; Colorectal Adenocarcinoma; Metastatic Solid Tumor; Recurrent Solid Tumor; Head and Neck Cancer
Keywords: NT219; ERBITUX; Cetuximab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation of NT219 as a single agent (Experimental)
  Interventions: Drug: NT219
- Dose escalation of NT219 in combination with ERBITUX® (Experimental)
  Interventions: Drug: NT219 and ERBITUX® - Dose Escalation
- Expansion cohort of NT219 in combination with ERBITUX® (Experimental)
  Interventions: Drug: NT219 and ERBITUX® - Expansion

INTERVENTIONS:
Drug: NT219 — Dose escalation of NT219 as a single agent in adult subjects with recurrent and/or metastatic solid tumors
  Arms: Dose escalation of NT219 as a single agent
Drug: NT219 and ERBITUX® - Dose Escalation — Dose escalation of NT219 in combination with standard dose ERBITUX® in adult subjects with recurrent and/or metastatic squamous cell carcinoma of the head and neck and colorectal adenocarcinoma
  Arms: Dose escalation of NT219 in combination with ERBITUX®
Drug: NT219 and ERBITUX® - Expansion — Expansion cohort of NT219 at its RP2D in combination with standard dose ERBITUX® in adult patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck
  Arms: Expansion cohort of NT219 in combination with ERBITUX®

SUMMARY:
This is a phase 1/2, multi-center study with an open-label, dose escalation phase followed by a single-arm expansion phase to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of NT219 alone and in combination with ERBITUX® (cetuximab) in adults with recurrent and/or metastatic solid tumors.

ELIGIBILITY:
Portion #2: Dose escalation of NT219 in combination with ERBITUX® in adult subjects with recurrent and/or metastatic squamous cell carcinoma head and neck and colorectal adenocarcinoma Inclusion Criteria

1. Subject with previously treated colorectal or head and neck cancer with documentation of incurable locally advanced, recurrent and/or metastatic squamous cell carcinoma of the head and neck or colorectal adenocarcinoma, stage III/IV that must have failed or not be a candidate for available standard of care therapies and not deemed amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy) by a multidisciplinary committee to include an oncologist, surgeon, and radiation oncologist
2. Subjects with head and neck cancer should have received up to 2 previous regimens for recurrent/metastatic disease; Only subjects with documented wild-type KRAS and BRAF colorectal cancer are allowed to enroll; subjects with colorectal cancer should have received up to 3 previous regimens for metastatic disease.
3. Subjects with HPV negative status only to be enrolled (for subjects with head and neck cancer)
4. Completion of curative radiation therapy at least 4 weeks prior to study treatment initiation; For subjects with head and neck cancer - prior focal palliative radiotherapy must be completed at least 2 weeks prior to study drug administration
5. Availability of archival tumor samples prior to treatment initiation; When not available or feasible for any reason, this requirement can be waived after discussion with the Sponsor.
6. Fresh tumor biopsy should be obtained unless deemed by the investigator that the procedure may pose a risk of bleeding to the subject or otherwise deemed not medically safe and/or feasible for any reason. This biopsy must be either formalin-fixed, paraffin-embedded (FFPE) tissue block or unstained tumor tissue samples, obtained within 3 months prior to enrollment and after the last systemic treatment was completed, with an associated pathology report. Biopsy should be excisional, incisional or core needle. Fine needle aspiration biopsy of the involved neck lymph nodes is permitted however, fine needle aspiration or biopsies of bone lesions that do not have a soft tissue component are unacceptable for submission.
7. Must have at least 1 measurable lesion per RECIST1.1 with progressing or new lesions since last antitumor therapy.
8. Age ≥18 years at the time of signing ICF;
9. ECOG performance status score of <2 at Screening and Baseline (Day 0);
10. Adequate safety lab results at Screening and at Baseline (Day 0) for those tests that require repeating at Baseline, including the following:

    1. Albumin ≥3 g/dL
    2. Bilirubin ≤1.5 times the upper limit of normal (ULN) or <3 times the ULN in the case of Gilbert Syndrome
    3. Aspartate aminotransaminase (AST), alanine aminotransaminase (ALT), and alkaline phosphatase <3 times the ULN
    4. Creatinine clearance >60 mL/minute based on the Cockcroft-Gault equation [creatinine clearance in mL/min = (140 - age in years) x body weight (kg)/72 x serum creatinine (mg/dL); multiplied by 0.85 for women]
    5. White blood cell (WBC) count ≥2000/uL; hemoglobin ≥9 g/dL;
11. Brain metastases should be stable following radiosurgery with at least 4 weeks since the end of definitive therapy (i.e., radiotherapy)
12. Subjects must have a "wash out" period of at least 4 weeks prior to first study drug administration from all previous chemotherapy and/or experimental agents except for anti-PD-1 antibodies which must have a "wash out" period of at least 6 weeks prior to first study drug administration, and all adverse events (AEs) have either returned to baseline or stabilized at Grade 1 or less.
13. Subject can understand and sign the ICF, can communicate with the PI, and can understand and comply with the requirements of the protocol;
14. WCBP must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 0)
15. WCBP must agree to abstain from sex or use an adequate method of contraception* from the time of informed consent through 2 months after the last dose of NT219;
16. Males must abstain from sex with WCBP or use an adequate method of contraception* from the time of informed consent through 2 months after the last dose of study drug.

    * Adequate contraceptive methods include those with a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as some double barrier methods (condom with spermicide) in conjunction with use by the partner of an intrauterine device, diaphragm with spermicide, oral contraceptives, birth control patch or vaginal ring, or injectable or implanted contraceptives. Abstinence is acceptable only as true abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

A woman that is postmenopausal (≥2 years since last menstrual period) or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) is not considered a WCBP.

Portion #3: Expansion cohort of NT219 in combination with ERBITUX® in adult subjects with recurrent and/or metastatic squamous cell carcinoma head and neck Inclusion Criteria

1. Subject with previously treated head and neck cancer, with documentation of incurable locally advanced, recurrent and/or metastatic squamous cell carcinoma of the head and neck, stage III/IV and not deemed amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy) by a multidisciplinary committee to include an oncologist, surgeon, and radiation oncologist
2. Patient has received up to 2 previous regimens for recurrent/metastatic disease;
3. Subjects with HPV negative status only to be enrolled Completion of curative radiation therapy at least 4 weeks prior to study treatment initiation; prior focal palliative radiotherapy must be completed at least 2 weeks prior to study drug administration
4. Availability of archival tumor samples prior to treatment initiation; When not available or feasible for any reason, this requirement can be waived after discussion with the Sponsor.
5. Fresh tumor biopsy should be obtained unless deemed by the investigator that the procedure may pose a risk of bleeding to the subject or otherwise deemed not medically safe and/or feasible for any reason. This biopsy must be either formalin-fixed, paraffin-embedded (FFPE) tissue block or unstained tumor tissue samples, obtained within 3 months prior to enrollment and after the last systemic treatment was completed, with an associated pathology report. Biopsy should be excisional, incisional or core needle. Fine needle aspiration biopsy of the involved neck lymph nodes is permitted however, fine needle aspiration or biopsies of bone lesions that do not have a soft tissue component are unacceptable for submission.
6. Must have at least 1 measurable lesion per RECIST1.1 with progressing or new lesions since last antitumor therapy.
7. Age ≥18 years at the time of signing ICF;
8. ECOG performance status score of <2 at Screening and Baseline (Day 0);
9. Adequate safety lab results at Screening and at Baseline (Day 0) for those tests that require repeating at Baseline, including the following:

   1. Albumin ≥3 g/dL
   2. Bilirubin ≤1.5 times the upper limit of normal (ULN) or <3 times the ULN in the case of Gilbert Syndrome
   3. Aspartate aminotransaminase (AST), alanine aminotransaminase (ALT), and alkaline phosphatase <3 times the ULN
   4. Creatinine clearance >60 mL/minute based on the Cockcroft-Gault equation [creatinine clearance in mL/min = (140 - age in years) x body weight (kg)/72 x serum creatinine (mg/dL); multiplied by 0.85 for women]
   5. White blood cell (WBC) count ≥2000/uL; hemoglobin ≥9 g/dL
10. Brain metastases should be stable following radiosurgery with at least 4 weeks since the end of definitive therapy (i.e., radiotherapy)
11. Subjects must have a "wash out" period of at least 4 weeks prior to first study drug administration from all previous chemotherapy and/or experimental agents except for anti-PD-1 antibodies which must have a "wash out" period of at least 6 weeks prior to first study drug administration, and all adverse events (AEs) have either returned to baseline or stabilized at Grade 1 or less.
12. Subject can understand and sign the ICF, can communicate with the PI, and can understand and comply with the requirements of the protocol
13. WCBP must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 0)
14. WCBP must agree to abstain from sex or use an adequate method of contraception* from the time of informed consent through 2 months after the last dose of NT219;
15. Males must abstain from sex with WCBP or use an adequate method of contraception* from the time of informed consent through 2 months after the last dose of study drug.

    * Adequate contraceptive methods include those with a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as some double barrier methods (condom with spermicide) in conjunction with use by the partner of an intrauterine device, diaphragm with spermicide, oral contraceptives, birth control patch or vaginal ring, or injectable or implanted contraceptives. Abstinence is acceptable only as true abstinence: when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

A woman that is postmenopausal (≥2 years since last menstrual period) or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) is not considered a WCBP.

Exclusion Criteria for Study Portions #2 & #3:

The exclusion criteria for Study Portion #2 drug combination dose escalation and Study Portion#3, the expansion phases of the trial are identical. Subjects meeting any of the following exclusion criteria will not be enrolled in the trial:

1. Nasal, paranasal sinus, or nasopharyngeal carcinoma and mutated KRAS colorectal adenocarcinoma, aside from World Health Organization (WHO) Type I and II [keratinizing, non-Epstein-Barr virus (EBV) positive] nasopharyngeal carcinoma which will be allowed;
2. In Study Part 2: For subjects with HNSCC: Received more than 2 prior systemic regimens for their HNSCC; For subjects with CRC: Received more than 3 prior systemic regimens for their CRC; In Study Part 3: For subjects with HNSCC: Received more than 2 prior regimens for their recurrent/metastatic HNSCC
3. Received cetuximab as part of the most recent regimen and/or within the last 6 months prior to study registration
4. Any invasive cancer (other than non-melanoma skin cancer) different from the current disease within 3 years of Screening
5. Known hypersensitivity to ERBITUX® or other epidermal growth factor receptor (EGFR), Janus kinase (JAK), or signal transducer and activator of transcription (STAT) antagonists/inhibitors, or inactive ingredients of NT219 Injection.
6. Radiation or major surgery within 4 weeks prior to the first dose of NT219;
7. Treatment with another investigational therapy within 30 days or 5 half-lives of the drug prior to Screening, whichever is longer
8. Parenteral vitamin C administration and oral supplements containing vitamin C
9. History of weight loss >10% over the 2 months prior to Screening
10. Active, untreated central nervous system (CNS) metastases
11. Severely immunocompromised as defined by white blood cell (WBC) count <2000/mm3 and/or CD4+ lymphocyte count ≤200/mm3
12. Major surgery within 4 weeks of study administration;
13. Known allergy to tick bites or red meat, or known immunoglobulin E (IgE) antibodies directed against galactose-α-1,3-galactose
14. Any condition which, in the opinion of the PI, places the subject at unacceptable risk if he/she were to participate in the study
15. Clinically relevant serious co-morbid medical conditions including, but not limited to:

    1. Active infection
    2. History of long QT syndrome or corrected QT interval (QTc) or QT/QTc interval measured as prolonged at screening (>480 ms; using Fredericia's QT correction formula). Note: subjects who screen fail due to this criterion are not eligible to be re-screened;
    3. A history of additional risk factors for TdP including clinically significant prolonged electrolytes imbalance, left ventricular dysfunction and left ventricular hypertrophy, prolonged diarrhea, bradycardia < 60 bpm, past history of syncope or a family history of sudden death at age <40 years
    4. The use of concomitant medications that prolong the QT/QTc interval or experienced arrhythmias with use of agents known to induce TdP.
    5. Recent (within six months of Screening) New York Heart Association (NYHA) Class III or IV cardiac disease, myocardial infarction, or severe or unstable angina;
    6. History of serious arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications
    7. Global Initiative for Chronic Obstructive Lung Disease (GOLD) score ≥3 chronic obstructive or chronic restrictive pulmonary disease, pulmonary hypertension, or interstitial pneumonitis
    8. Active CNS disease including carcinomatous meningitis;
    9. Psychiatric illness/social situation that would limit compliance with study requirements; Prior organ allograft
    10. Subjects with active, known or suspected autoimmune disease. Subjects with the following are permitted to enroll: (subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid patients with a history of Grave's disease (subjects with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study drug), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
    11. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration except for adrenal replacement steroid doses >10 mg daily prednisone equivalent in the absence of active autoimmune disease. Note: Treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study drug is permitted.
    12. History of active or latent tuberculosis infection
    13. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) as follows:

    Subjects with HIV: detectable viral load and CD4 count below 200 cells/mm3; Subjects with HBV (HepBsAg+): serum HBV DNA polymerase chain reaction (PCR) that is above the limit of detection Subjects with HCV (Ab +): detectable HCV RNA by PCR
16. Pregnant or lactating women
17. Use of UGT inhibitors within 14 days prior to first dose of study treatment. Morphine and similar agents and statins which are commonly used in oncology subjects are permitted. See Appendix E for sample list of prohibited UGT inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of treatment emergent adverse events | Up to 24 months
  Incidence of treatment emergent adverse events with single agent NT219
Part 2: Incidence of treatment emergent adverse events | Up to 24 months
  Incidence of treatment emergent adverse events with NT219 administered in combination with ERBITUX®
Part 3: Objective Response Rate | Up to 24 months
  Objective Response Rate when phase 2 dose of NT219 is used in combination with ERBITUX® in adults with recurrent and/or metastatic SCCHN

SECONDARY OUTCOMES:
Area under the plasma concentration curve [AUC] | Up to 45 days after first study drug administration
  Area under the plasma concentration curve [AUC] of NT219
Maximum plasma concentration [Cmax] | Up to 45 days after first study drug administration
  Maximum plasma concentration [Cmax] of NT219
Volume of distribution at stead-state [Vss] | Up to 45 days after first study drug administration
  Volume of distribution at stead-state [Vss] of NT219
Plasma half-life [t1/2] | Up to 45 days after first study drug administration
  Plasma half-life [t1/2] of NT219
Plasma clearance [Cl] | Up to 45 days after first study drug administration
  Plasma clearance [Cl] of NT219
Objective Response Rate when NT219 is used as monotherapy | Up to 24 months
Duration of Response when NT219 is used as monotherapy | Up to 24 months
Time to Response when NT219 is used as monotherapy | Up to 24 months
Disease Control Rate when NT219 is used as monotherapy | Up to 24 months
Progression Free Survival when NT219 is used as monotherapy | Up to 24 months
Time to Progression when NT219 is used as monotherapy | Up to 24 months
Overall Survival when NT219 is used as monotherapy | Up to 24 months
Objective Response Rate when NT219 is used in combination with ERBITUX® | Up to 24 months
Duration of Response when NT219 is used in combination with ERBITUX® | Up to 24 months
Time to Response when NT219 is used in combination with ERBITUX® | Up to 24 months
Disease Control Rate when NT219 is used in combination with ERBITUX® | Up to 24 months
Progression Free Survival when NT219 is used in combination with ERBITUX® | Up to 24 months
Time to Progression when NT219 is used in combination with ERBITUX® | Up to 24 months
Overall Survival when NT219 is used in combination with ERBITUX® | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schickler, PhD, Study Director — TyrNovo Ltd.
Locations (10):
- United States (7):
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - UCSD Moores Cancer Center, San Diego, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - The University of Chicago and Biological Sciences, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
- Israel (3):
  - Hadassah University Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No